CLINICAL TRIAL: NCT02712879
Title: Bleeding Moderate Postoperative Cardiac Surgery and Prognostic Implications Anemia and Postoperative Transfusion: Prospective, Observational, Descriptive.
Brief Title: Moderate Bleeding in Cardiac Surgery Post Operative
Acronym: SPO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF9695
Record Dates: First submitted 2016-03-04; First posted 2016-03-18 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Heart Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Determine a bleeding threshold by measuring the blood volume in ml / kg / h collected in the drainage system to define moderate bleeding postoperative cardiac surgery and define the population.

DETAILED DESCRIPTION:
Determine a bleeding threshold by measuring the blood volume in ml / kg / h collected in the drainage system to define moderate bleeding postoperative cardiac surgery and define the population.

Secondary objectives:

To evaluate the kinetics of moderate SPORT and its impact on anemia and postoperative transfusion.

To evaluate the prognostic impact of the SPO moderate in terms of post-operative complications.

Determine predictors of moderate SPO.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the postoperative intensive care in cardiac surgery

Exclusion Criteria:

* Patients who received a heart transplant, a heart surgery beating, cardiac support establishment of long duration, or have a disease that alters the coagulation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to intensive care after surgery for heart surgery
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Evolution of blood loss per hour drains | Hourly blood loss in drains during the first twelve hours
  Hourly blood loss in drains during the first twelve hours

CONTACTS AND LOCATIONS:
Overall Officials: Marine SAOUR, CCA, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UHMontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided